CLINICAL TRIAL: NCT00898976
Title: Molecular Markers in Native American Women With Breast Cancer
Brief Title: Biomarkers in Native American Women With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCCTG-97-95-51; NCCTG-979551; CDR0000078596 (Registry Identifier: PDQ (Physician Data Query)); NCI-2013-00323 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; breast cancer in situ; recurrent breast cancer; stage IIIB breast cancer; inflammatory breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Inflammatory Breast Neoplasms | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group I: Immunohistochemistry is performed on tumor samples to analyze the following molecular markers: estrogen receptor, progesterone receptor, c-erbB2, p53, Ki-67, Bcl-2, Bax, cyclin D-1, and insulin-like growth factor-1R. PROJECTED ACCRUAL: A total of 300 tissue samples (150 from Native American women and 150 from Caucasian women) will be accrued for this study.
  Interventions: Other: immunohistochemistry staining method; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue in the laboratory from Native American women with breast cancer may help doctors identify and learn more about biomarkers related to breast cancer in these patients. It may also help doctors learn more about the prognosis of these patients.

PURPOSE: This laboratory study is looking at biomarkers in Native American women with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate a selected panel of molecular markers in tissue specimens from Native American women with breast cancer.
* Determine which molecular markers provide independent prognostic information with respect to traditional prognostic factors in these patients.
* Compare and contrast the prevalence of positivity in Native American women with breast cancer with an age- and stage-matched cohort of Caucasian women with breast cancer enrolled on clinical trial NCCTG-77-30-51 or the Mayo Breast Cancer Registry.

OUTLINE: Immunohistochemistry is performed on tumor samples to analyze the following molecular markers: estrogen receptor, progesterone receptor, c-erbB2, p53, Ki-67, Bcl-2, Bax, cyclin D-1, and insulin-like growth factor-1R.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary adenocarcinoma of the breast in Native American women
* Prior surgical treatment for breast cancer within the Aberdeen or Phoenix areas of the Indian Health Service or the Alaska area of the Native Health Service between 1990-2000

  * Paraffin-embedded tissue available
* Paraffin-embedded tissue available from Caucasian women with breast cancer enrolled on NCCTG-77-30-51 or the Mayo Breast Cancer Registry

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Native American women with primary adenocarcinoma of the breast with prior surgical treatment for breast cancer within the Aberdeen or Phoenix areas of the Indian Health Service or the Alaska area of the Native Health Service between 1990-2000.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 1998-08; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of a selected panel of molecular markers in tissue specimens from Native American women with breast cancer | Up to 5 years
Determination of which molecular markers provide independent prognostic information with respect to traditional prognostic factors | Up to 5 years
Comparison of the prevalence of positivity in Native American women with breast cancer with an age- and stage-matched cohort of Caucasian women with breast cancer enrolled on clinical trial NCCTG-77-30-51 or the Mayo Breast Cancer Registry | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Judith S. Kaur, MD, Study Chair — Mayo Clinic